CLINICAL TRIAL: NCT02466061
Title: Transdisciplinary Research on Energetics (TREC) and Cancer Cross Center Study / Obesity and Weight Loss in Endometrial Cancer Survivors: A Randomized, Multi-site Trial (Lifestyle Beyond Cancer Study)
Brief Title: TREC Lifestyle Beyond Cancer Study in Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Pennsylvania (Other); Washington University School of Medicine (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: TREC 1190; U01CA116850 (NIH); U54CA155850 (NIH); U54CA155496 (NIH); U54CA155626 (NIH)
Record Dates: First submitted 2015-05-29; First posted 2015-06-09 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Endometrial Cancer
Keywords: BMI >= 30 kg/m2
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Diet; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: Telemedicine Group (Experimental): Telemedicine Weight Management plus Wi-Fi Scale (Arm A) Participants in the Telemedicine Group will receive a Wi-Fi Scale that measures weight, lean mass, and fat mass. Participants will receive 15-20 minute telephone counseling sessions by phone. Sessions will occur at routine intervals during the six month intervention period.
  All Aim 1 participants, including those randomized to Arm A, will complete a packet of psychosocial measures at baseline and 6 months (final assessment).
  Month 12 followup weight data also will be collected through medical record abstraction.
  Interventions: Behavioral: Telemedicine Weight Management plus Wi-Fi Scale (Arm A)
- Arm B: Text for Diet (Text4Diet) Group (Experimental): Text for Diet (Text4Diet) Group (Arm B) The intervention in this Arm involves delivery of Short Message Service (SMS) text messages to participants each day over the course of a 6 month intervention period. Participants will also receive a digital scale to track weight on a weekly basis. SMS text messages will be sent 2-3 times per day and will provide feedback, support, prompting, and strategies to adhere to behaviors associated with long-term weight management.
  All Aim 1 participants, including those randomized to Arm B, will complete a packet of psychosocial measures at baseline and 6 months (final assessment).
  Month 12 follow up weight data also will be collected through medical record abstraction.
  Interventions: Behavioral: Text for Diet (Text4Diet) Group (Arm B)
- Arm C: Enhanced Usual Care Group (Active Comparator): Enhanced Usual Care Group (Arm C) Participants will be provided with handouts based on American Cancer Society guidelines on healthy eating and exercise.
  All Aim 1 participants, including those randomized to Arm C, will complete a packet of psychosocial measures at baseline and 6 months (final assessment).
  Month 12 follow up weight data also will be collected through medical record abstraction.
  Interventions: Behavioral: Enhanced Usual Care Group (Arm C)

INTERVENTIONS:
Behavioral: Telemedicine Weight Management plus Wi-Fi Scale (Arm A) — Telephonic weight loss counseling by trained interventionists, with guided digital scale measurements of weight, lean mass, and fat mass. Counseling sessions and digital weight recording occur at regularly scheduled intervals over a six-month intervention period.
  Other Names: Telemedicine Group
  Arms: Arm A: Telemedicine Group
Behavioral: Text for Diet (Text4Diet) Group (Arm B) — Short Message Service (SMS) text messaging in which participants receive 3-5 text messages each day during a six-month intervention period. The text messages provide tips and reminders to encourage healthy eating and weight loss. Participants on this arm also receive a digital scale to track and report weight as prompted once per week through the text program.
  Other Names: Text4Diet Group
  Arms: Arm B: Text for Diet (Text4Diet) Group
Behavioral: Enhanced Usual Care Group (Arm C) — Participants are provided with handouts based on American Cancer Society guidelines for healthy eating and exercise.
  Other Names: Enhanced Usual Care Group
  Arms: Arm C: Enhanced Usual Care Group

SUMMARY:
This randomized, controlled study evaluates the efficacy of weigh loss interventions in endometrial cancer survivors, using novel technology-based weight loss platforms. This is a multi-site, pilot feasibility study which will provide preliminary data to support a larger NIH funded, mult-center trial.

DETAILED DESCRIPTION:
Study Aims The relationship between endometrial cancer (EC) and obesity is well established. However, few studies have examined the acceptability and potential efficacy of an intervention to promote weight reduction and alter cancer-associated biomarkers in endometrial cancer survivors. This investigation has two specific aims.

Aim 1:

To compare the efficacy of novel technology-based weight loss interventions: a) telephone encounters and wireless scales, or b) smart phone personalized text messaging as compared to c) an enhanced usual care group for women with obesity and a history of endometrial cancer.

Hypothesis: Women in both the telemedicine and text intervention arms will lose significantly more weight than women in the enhanced usual care arm.

Aim 2:

1a) To explore patients' understanding of the relationship between obesity and endometrial cancer and, 1b) to survey the acceptability of novel and different approaches to weight loss.

Hypothesis: The investigators anticipate that this study will validate pilot data from a predecessor single-institution study demonstrating that >25% of patients will not be aware of the association between excess body weight and endometrial cancer. Investigators also will assess the acceptability of various interventions designed to promote weight loss (i.e. in person counseling, phone-based, text messaging) and predict a greater interest in interventions that require fewer in-person visits to the clinic.

Study Design

Aim 1:

* 3 arm randomized controlled trial, weight loss intervention
* Pre and post intervention patient reported psychosocial measures
* Pre and post intervention Dual-energy X-ray absorptiometry (DEXA) to explore impact of weight loss on body fat distribution
* Pre and post intervention analyses of the following biomarkers: insulin-like growth factor-binding protein 1 (IGFBP-1); adiponectin, vascular endothelial growth factor (VEGF), C reactive protein (CRP), interleukin 1-beta (IL1-beta), interleukin 2 (IL2), interleukin 6 (IL6), interleukin 7 (IL7), and interleukin 8 (IL8)

Aim 2: Patient-reported survey to assess knowledge of correlation of Body Mass Index (BMI) with endometrial cancer incidence

Study Population

Aim 2: Adult women with biopsy-proven endometrial cancer (Types I and II), BMI ≥ 30 kg/m2.

Aim 1: Aim 2 population plus Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1, no concurrent chemo or radiation therapy, and access to wireless internet and/or smart phone device.

ELIGIBILITY:
Inclusion Criteria:

Aim 2

1. Women 18 years of age or older and with biopsy-proven endometrial cancer,
2. Body Mass Index (BMI) greater than or equal to 30 kg/m2 (based on most recent routine clinical measurement recorded in patient's medical record),
3. Must be able to read and speak English fluently, and
4. All patients must be informed of the investigational nature of the Aim 2 survey study and must give written informed consent for Aim 2 study activities in accordance with institutional and federal guidelines. (Aim 2 consent is obtained and documented as described on page 1 of the Endometrial Cancer Questionnaire).

Aim 1

1. Woman who was recruited to and completed Aim 2 of the study,
2. Has completed prior surgical or other medical management and adjuvant endometrial cancer treatment, prior to starting Aim 1,
3. Is not receiving concurrent cytotoxic chemotherapy and/or radiation therapy at time of randomization AND, after randomization, it is not anticipated that the participant will need to receive concurrent cytotoxic chemotherapy and/or radiation therapy at any time during the Aim 1 intervention,
4. No evidence of active endometrial cancer disease as determined by physician evaluation prior to randomization,
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
6. Life expectancy of at least one year,
7. Must have access to either wireless Internet, or a smart phone such as an Android or Apple iPhone, and
8. All patients must be informed of the investigational nature of this study and must sign and give written informed consent for Aim 1 study activities in accordance with institutional and federal guidelines.

Exclusion Criteria:

Aim 2

1. Must not have any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with Aim 2 protocol compliance or a participant's ability to give informed consent.

   4.3.2.2 Aim 1
2. Must not be participating in another weight loss program or taking weight loss medications,
3. No uncontrolled serious medical or psychiatric condition(s) that would affect the patient's ability to participate in the interventional study, e.g., uncontrolled hypertension, symptomatic cardiac disease, or severe/uncontrolled depression as indicated by a Patient Health Questionnaire (PHQ-9) score >19, or a score of ≥1 on the suicidal ideation item (#9 on the PHQ-9)
4. No diagnoses of any other invasive malignancy other than endometrial cancer or non-melanoma skin cancer which required active treatment currently or within the last 5 years. Carcinosarcoma is not excluded as the investigators are including women with Type I and II endometrial cancer. For the purposes of the trial, carcinosarcoma falls into the Type II category.
5. No diagnoses of autoimmune disorders (including lupus, rheumatoid arthritis, Siogren's syndrome, Crohn's disease and ulcerative colitis), immune-compromised disorders (i.e., HIV/AIDS),
6. Not receiving at time of randomization, and not expected to receive at any time during the Aim 1 intervention, any medications that may affect the inflammatory markers of interest (i.e., steroids, immunosuppressants or transplant medications), and
7. Must not have any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with Aim 1 protocol compliance or a participant's ability to give informed consent.
8. Must not be pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Weight (kilograms) | Change from Baseline Weight at 6 months
  Change in weight (in kilograms) of study participants randomized to one of three weight loss intervention programs will be assessed. Measurement of this change will be evaluated from weights taken at baseline (randomization) and six months, the conclusion of the intervention program.
Serum biomarker: Change in levels of Insulin-like growth factor-binding protein 1 (IGFBP-1), in ng/mL | Change from Baseline IGFBP-1 at 6 months
  Change in IGFBP-1 (in ng/mL) of randomized study participants will be assessed in peripheral blood samples collected at baseline (randomization) and again at 6 months, the conclusion of the intervention program.
Serum biomarker: Change in levels of Adiponectin, in ug/mL | Change from Baseline Adiponectin at 6 months
  Change in Adiponectin (in ug/mL) of randomized study participants will be assessed in peripheral blood samples collected at baseline (randomization) and again at 6 months, the conclusion of the intervention program.
Serum biomarker: Change in levels of Vascular Endothelial Growth Factor (VEGF), in pg/mL | Change from Baseline VEGF at 6 months
  Change in VEGF (in pg/mL) of randomized study participants will be assessed in peripheral blood samples collected at baseline (randomization) and again at 6 months, the conclusion of the intervention program.
Serum biomarker: Change in Interleukin 1-beta (IL1-beta), in pg/mL | Change from Baseline IL1-beta at 6 months
  Change in IL1-beta (in pg/mL) of randomized study participants will be assessed in peripheral blood samples collected at baseline (randomization) and again at 6 months, the conclusion of the intervention program.
Serum biomarker: Change in Interleukin 2 (IL2), in pg/mL | Change from Baseline IL2 at 6 months
  Change in IL2 (in pg/mL) of randomized study participants will be assessed in peripheral blood samples collected at baseline (randomization) and again at 6 months, the conclusion of the intervention program.
Serum biomarker: Change in Interleukin 6 (IL6), in pg/mL | Change from Baseline IL6 at 6 months
  Change in IL6 (in pg/mL) of randomized study participants will be assessed in peripheral blood samples collected at baseline (randomization) and again at 6 months, the conclusion of the intervention program.
Serum biomarker: Change in Interleukin 7 (IL7), in pg/mL | Change from Baseline IL7 at 6 months
  Change in IL7 (in pg/mL) of randomized study participants will be assessed in peripheral blood samples collected at baseline (randomization) and again at 6 months, the conclusion of the intervention program.
Serum biomarker: Change in Interleukin 8 (IL8), in pg/mL | Change from Baseline IL8 at 6 months
  Change in IL8 (in pg/mL) of randomized study participants will be assessed in peripheral blood samples collected at baseline (randomization) and again at 6 months, the conclusion of the intervention program.
Serum biomarker: Change in C reactive protein (CRP), in mg/L | Change from Baseline CRP at 6 months
  Change in CRP (in mg/L) of randomized study participants will be assessed in peripheral blood samples collected at baseline (randomization) and again at 6 months, the conclusion of the intervention program.

SECONDARY OUTCOMES:
Knowledge of the association between obesity and endometrial cancer risk | Baseline
  Participants' level of knowledge of the association between obesity and the risk of endometrial cancer will be assessed at baseline. Frequencies of categorical responses will be reported. The instrument used to collect this data is a participant completed Endometrial Cancer Questionnaire and was developed by the study investigators.
Psychosocial measure: Change in Body Image | Change from Baseline Body Image at 6 months
  Change in participants' self-reported body image will be assessed at baseline (randomization) and again at 6 months, the conclusion of the intervention program. Two validated, participant-completed instruments will be utilized to assess this outcome: the Multidimensional Body Self Relations Questionnaire-Appearance Subscales (MBSRQ-AS) and the Cancer-Related Body Image Scale (CRBI).
Psychosocial measure: Change in Quality of Life | Change from Baseline in Quality of Life at 6 months
  Change in participants' self-reported quality of life will be assessed at baseline (randomization) and again at 6 months, the conclusion of the intervention program. One validated, participant-completed instrument will be utilized to assess this outcome: the 12-Item Short Form Health Survey (SF-12).
Psychosocial measure: Change in Mood | Change from Baseline in Mood at 6 months
  Change in participants' self-reported quality of life will be assessed at baseline (randomization) and again at 6 months, the conclusion of the intervention program. One validated, participant-completed instrument will be utilized to assess this outcome: the Patient Health Questionnaire 9-Item Version (PHQ-9).
Psychosocial measure: Change in Sexual Functioning | Change from Baseline in Sexual Functioning at 6 months
  Change in participants' self-reported sexual functioning will be assessed at baseline (randomization) and again at 6 months, the conclusion of the intervention program. Three validated, participant-completed instruments will be utilized to assess this outcome: the Female Sexual Function Index (FSFI), the Dyadic Adjustment Scale (DAS), and the Female Sexual Distress Scale-Revised (FSDS-R).
Psychosocial measure: Change in Physical Activity | Change from Baseline Physical Activity at 6 months
  Change in participants' self-reported physical activity will be assessed at baseline (randomization) and again at 6 months, the conclusion of the intervention program. One validated, participant-completed instrument will be utilized to assess this outcome: the International Physical Activity Questionnaire Short Form (IPAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Allison, PhD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University in St Louis (Siteman Cancer Center), St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Haggerty AF, Hagemann A, Barnett M, Thornquist M, Neuhouser ML, Horowitz N, Colditz GA, Sarwer DB, Ko EM, Allison KC. A Randomized, Controlled, Multicenter Study of Technology-Based Weight Loss Interventions among Endometrial Cancer Survivors. Obesity (Silver Spring). 2017 Nov;25 Suppl 2(Suppl 2):S102-S108. doi: 10.1002/oby.22021. PMID 29086522